CLINICAL TRIAL: NCT03081806
Title: A Phase 3, Multicenter, Randomized, Placebo-controlled, Double-blind, 22-Week and 30-Week Open-label Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of X0002 Spray in Relief of the Pain for Subjects With Osteoarthritis of the Knee
Brief Title: A Study to Evaluate the Efficacy and Safety of X0002 Spray in Subjects With Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Techfields Pharma Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TF-X0002-31
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Pain Associated With Osteoarthritis of the Knee
Keywords: Phase 3; Efficacy; Safety; Osteoarthritis, Knee, Pain
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): High dose group: X0002, BID (approximately every 12 hours; n=102); Placebo, BID(approximately every 12 hours; n=102)
  Interventions: Drug: X0002
- Group B (Placebo Comparator): Low dose group: X0002, BID (approximately every 12 hours; n=102); Placebo, BID(approximately every 12 hours; n=102)
  Interventions: Drug: X0002

INTERVENTIONS:
Drug: X0002 — Subjects will complete 22 weeks of double-blind treatment and then enter into 30 weeks open-label treatment.

SUMMARY:
This is a Phase 3, Multicenter, 22-Week, double-blind and 30-Week open label Study to Evaluate the Efficacy and Safety of X0002 Spray in relief of pain of subjects with Osteoarthritis of the Knee.

DETAILED DESCRIPTION:
The study comprises a 14-day Screening Period, a 22-week Double-blind Treatment Period, and a 30-week Open-label Treatment Period, with an additional 4-week Follow-up Visit. Subjects will be randomized into a low-dose or high-dose group receiving either active or placebo treatment during the DB period.

The WOMAC version 3.1 using the NRS will be used for the primary and secondary efficacy endpoints. Safety assessments will include assessment of AEs, vital signs (blood pressure, respiratory rate, pulse rate, and oral temperature), clinical laboratory tests, physical examination, skin irritation, and electrocardiograms (ECGs).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to read and provide written, personally signed, and dated informed consent to participate in the study, in accordance with the ICH GCP Guideline E6 and applicable regulations, before completing any study related procedures.
2. An understanding, ability, and willingness to fully comply with study procedures and restrictions.
3. Subject must be a male or female between 35 and 85 years of age, inclusive.
4. Female subjects must either not be of childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) or be willing to Practice at least 1 of the following medically acceptable methods of birth control.
5. Subject must have a body mass index (BMI) between 18.5 and 45 kg/m2, inclusive.
6. Must have a history of clinically symptomatic OA of the knee for ≥6 months.
7. Must meet the American College of Rheumatology clinical classification criteria for knee OA. These criteria include the presence of knee pain in addition to at least 3 of the following 6 items:

   * age of ≥50 years
   * stiffness lasting <30 minutes
   * crepitus on knee motion
   * Bony Tenderness
   * Bony Enlargement
   * No palpable warmth
8. A subject must have a Kellgren Lawrence Grade of 2,3 or 4 as determined by a central radiologist at the first screening visit. .
9. Subject must have had knee pain while standing, walking, and/or in motion for at least 14 days during the month prior to Screening.
10. Subject must have a knee pain score ≥4 and <9 on 0-10 pain intensity NRS (without analgesic medication) on at least 7 of the 10 days prior to randomization.
11. Subject must be willing to discontinue any NSAIDs or other analgesic (eg, aspirin, acetaminophen) or potentially confounding concomitant treatments (eg, physiotherapy, acupuncture) starting on the first screening visit until completing participation in the study. (The use of ≤325 mg acetylsalicylic acid per day as cardiac prophylaxis is permitted.) The subject will be allowed to take rescue medication (acetaminophen) for pain during the study except during the 24 hours prior to the Second Screening Visit, Baseline (Day1), Week 2, Week 4, Week 8, Week 12, Week 22, Week 32, Week 42, and Week 52/EOS.
12. Subject must be willing to discontinue applying any topical preparations containing Vitamin A acids (including all trans retinoic acid (tretinoin), 13 cis retinoic acid [isotretinoin], 9 cis retinoic acid [alitretinoin], vitamin A [retinol], retinal, and their derivatives) to the lower limbs starting on the first screening visit until completing participation in the study. (Topical preparations containing Vitamin A acids or retinol may be applied to areas of the skin above the waist, but should not be applied to areas of the skin exposed to study medication.)
13. Subject must be willing to avoid unaccustomed physical activity (eg, starting a new weight lifting routine) for the duration of the study starting on the first screening visit.
14. With the exception of OA of the knee subjects with medical history must be stable as determined by the investigator.

Exclusion Criteria:

1. Has worker's compensation injuries affecting the knee or back.
2. Has a history of or is currently in litigation regarding joint injuries.
3. Has secondary OA of the target knee or OA of lower limb joints other than the knee that, in the investigator's opinion, could interfere with pain and functional assessments related to the target knee.
4. Has a history of total or partial knee replacement, arthroplasty, or other knee surgery on the target knee.
5. In the investigator's opinion, has had significant injury involving the target knee within the 6 months before Screening.
6. Has skin lesions or wounds on or near the target knee at Screening or at Baseline (Day 1) that, in the investigator's opinion, would affect absorption of the medication.
7. Has used opiates (including tramadol or tapentadol) or systemic corticosteroids within 30 days before Screening or requires treatment with chronic opiates or systemic corticosteroids.
8. Subjects with a placebo response exceeding 25% improvement in the average Western Ontario and McMaster Osteoarthritis Index [WOMAC] pain subscale score from Screening Visit to Day 1 will be excluded.
9. Has used gabapentin, pregabalin, antiepileptics, or specific antidepressants (i.e., tricyclics, serotonin norepinephrine reuptake inhibitors, or selective serotonin reuptake inhibitors) to treat pain in the 14 days before Screening. Other uses not related to the pain treatment may be permitted at the medical monitor's discretion provided they have been at a stable dose for at least 90 days.
10. Has had intra articular (IA) injections of corticosteroids, hyaluronic acid, or viscosupplements (e.g., Synvisc®) to the target knee within the 12 weeks before Screening
11. Has had IA or intravenous (IV) stem cell therapy in the 6 months prior to Screening
12. Is receiving or is planning to receive concomitant nonpharmacologic treatments (e.g., physiotherapy, acupuncture) that in the investigator's opinion could confound efficacy assessments within 14 days of Day 1.
13. Has a history of significant hypersensitivity, intolerance, or allergy to ibuprofen or any other NSAIDs, aspirin, or acetaminophen.
14. Has had an active gastrointestinal (GI) ulceration in the 6 months prior to Screening or a history of GI bleeding within 5 years of Screening.
15. Has used an anticoagulant or antiplatelet agent (except aspirin up to 325 mg/day for cardiac prophylaxis) in the 30 days prior to Screening.
16. Has a documented history of chronic inflammatory disease (e.g., rheumatoid arthritis, psoriatic arthritis, inflammatory bowel disease, gouty arthritis) OR chronic pain condition (e.g., fibromyalgia), OR has other conditions that may affect the target joint for the functional and pain assessments (e.g., osteonecrosis, chondrocalcinosis).
17. Has uncontrolled depression or other uncontrolled psychiatric disorder (subjects with controlled depression or other psychiatric disorder, if using medication, must be on a stable dose of a medication other than an epileptic, tricyclic, serotonin norepinephrine reuptake inhibitor, or selective reuptake inhibitor for ≥12 weeks prior to Screening to participate in the study).
18. Has asthma requiring treatment with systemic corticosteroids in the last year prior to Screening. Asthmatic subjects using inhaled corticosteroids are eligible.
19. Has uncontrolled hypertension defined as systolic blood pressure >170 mmHg and diastolic blood pressure >90 mmHg at the Screening or Baseline Visit (may be repeated after 5 minutes rest to verify).
20. Is receiving systemic chemotherapy, has an active malignancy, lymphoproliferative disorder, or blood dyscrasia of any type, or has been diagnosed with cancer within 5 years before Screening. Subjects with completely excised squamous or basal cell carcinoma of the skin will be allowed.
21. Has any clinically significant unstable cardiac, respiratory, neurological, immunological, hematological, hepatic, or renal disease, or any other condition that, in the Investigator's opinion, could confound the study results, compromise the subject's welfare, interfere with the ability to communicate with the study staff, or otherwise contraindicate study participation.
22. Has any of the following conditions at Screening:

    * Acute hepatitis
    * Cirrhosis
    * Stage 4 or 5 end-stage renal disease
23. Subject has any other clinically significant laboratory finding at Screening that in the investigator's opinion contraindicates study participation.
24. Has clinically significant abnormality at Screening or Baseline (Day 1) on 12-lead ECG, including a QT interval calculated using Fridericia's correction (QTcF) interval >500 milliseconds (msec) or evidence of cardiac ischemia (i.e., Evident q waves: t wave inversion).
25. Is pregnant, planning to become pregnant during the study, or lactating. Has a positive serum and urine pregnancy test at Screening Visit, or a positive urine pregnancy test at Baseline (Day 1).
26. Has a positive urine drug screen for a nonprescribed drug prohibited by the protocol at Screening.
27. Has known alcohol or other substance abuse in the investigator's opinion.
28. Has participated in a previous clinical study with X0002.
29. Has participated in any other clinical trial within the past 30 days or within 5 half-lives of the study drug prior to Screening, whichever is longer.
30. Is a participating investigator, sub-investigator, study coordinator, or employee of a participating investigator, or is an immediate family member of the aforementioned.
31. Has any factor that, in the investigator's opinion, would jeopardize the evaluation or safety or be associated with poor adherence to the protocol.
32. Is without access to telephone and/or ability to gain technology access.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
WOMAC pain subscale score in the target knee at Week 12 compared to Baseline | Week 12
  To evaluate the effect of X0002 spray compared to placebo for relief of knee pain in subjects with OA of the knee as measured by the WOMAC pain subscale score in the target knee at Week 12.

SECONDARY OUTCOMES:
Subject's Global Assessment of Disease Status at Week 12. | Week 12 of treatment
  To evaluate the effect of X0002 spray for Subject's Global Assessment of Disease Status in subjects with OA of the knee in the target knee.
WOMAC fuctional subscale score in the target knee at Week 12 | Week 12 of treatment
  To evaluate the effect of X0002 spray for relief of fuctional subscale in subjects with OA of the knee as measured by the WOMAC pain subscale score in the target knee at Week 12.
WOMAC (NRS) pain subscale in the target knee at Week 2, 4, 8, and 22 | Week 2, 4, 8 , and 22 of treatment
  To evaluate the efficacy of X0002 spray in average WOMAC (NRS) pain subscale in the target knee at Weeks 2, 4, 8, and 22
WOMAC function subscale score | Week 2, 4, 8 , and 22 of treatment
  To evaluate the efficacy of X0002 spray in changes of WOMAC function subscale score of subjects with osteoarthritis (OA) of the target knee at Week 2, 4, 8 and 22.
Average eDiary daily (NRS) score in the target knee | Week 2, 4, 8, 12 and 22 of treatment
  To evaluate the change from Baseline in average eDiary daily (NRS) score in the target knee for the 7 days prior to Weeks 2, 4, 8, 12, and 22.
WOMAC overall score | Week 2, 4, 8, 12 and 22 of treatment
  To evaluate the efficacy of X0002 spray in change WOMAC overall score of subjects with osteoarthritis (OA) of the target knee at Weeks 2, 4,8,12 and 22.
WOMAC stiffness subscale | Week 2, 4, 8, 12 and 22 of treatment
  To evaluate the efficacy of X0002 spray in change WOMAC stiffness subscale of subjects with osteoarthritis (OA) of the target knee at Weeks 2, 4,8,12 and 22.

CONTACTS AND LOCATIONS:
Overall Officials: Chongxi Yu, PhD, Study Chair — Techfields Inc
Locations (33):
- United States (33):
  - Arizona Research Center, Phoenix, Arizona
  - Yuma Clinical Trials, Yuma, Arizona
  - Orange County Research Institute, Anaheim, California
  - Biosolutions Clinical Research Center, La Mesa, California
  - Velocity Clinical Research, North Hollywood, California
  - University Clinical Research-Deland, DeLand, Florida
  - Reliable Clinical Research, Hialeah, Florida
  - Health Awareness Inc., Jupiter, Florida
  - Ascension Research, Pinellas Park, Florida
  - Conquest Research, Winter Park, Florida
  - Horizon Clinical Research, Newnan, Georgia
  - Pinnacle Trials Inc, Stockbridge, Georgia
  - Chicago Clinical Research Institute Inc, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Healthcare Research Network, Flossmoor, Illinois
  - Affinity Health Corp, Oak Brook, Illinois
  - DelRicht Research, New Orleans, Louisiana
  - DelRicht Research, Prairieville, Louisiana
  - DelRicht Research - Gulfport, Gulfport, Mississippi
  - Healthcare Research Network, LLC, Hazelwood, Missouri
  - AMR Kansas City, Kansas City, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - AMR: Las Vegas, Las Vegas, Nevada
  - Upstate Clinical Research Associates LLC, Williamsville, New York
  - Aventiv Research, Inc - Brice Road Location, Columbus, Ohio
  - DelRicht Research, Tulsa, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Tekton Research, Austin, Texas
  - Clinical Investigations of Texas, Plano, Texas
  - Quality Research Inc., San Antonio, Texas
  - Wasatch Clinical Research LLC, Salt Lake City, Utah
  - Charlottesville Medical Research, LLC, Charlottesville, Virginia
  - Spectrum Medical, Inc, Danville, Virginia

IPD SHARING:
Plan to Share IPD: No